CLINICAL TRIAL: NCT02508818
Title: Cardiovascular Response to Orthostatic Fractional Gravity
Acronym: ORB
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 11-010
Record Dates: First submitted 2015-07-23; First posted 2015-07-27 (Estimated); Last update posted 2015-07-27 (Estimated); Status verified 2015-07

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cardiovascular measurements (Other)
  Interventions: Other: Parabolic flight; Other: Cardiovascular measurements

INTERVENTIONS:
Other: Parabolic flight
Other: Cardiovascular measurements

SUMMARY:
There are no equivalent experiment setups to create comparable changes of gravitation such as during parabolic flights. To determine the initial orthostatic responses of the cardiovascular system under the gravitational conditions of mars and moon is an essential step for a better understanding of 1) the fundamental functions of the human cardiovascular system (basic research) 2) specific impact of partial-g on the human heart, lungs and vessels in a spaceflight-context 3) approaches for countermeasure development against orthostatic intolerance on moon and mars (applied research).

Non-invasive measurement methods will be used to achieve the cardiovascular key values of the study: stroke volume (SV) and cardiac output determination by pulse contour analysis, impedance cardiography and inert gas rebreathing, beat-to-beat finger blood pressure measurement, heart rate and heart rate variability determination by ECG. All of these methods have proven their accuracy during parabolic flights. Nevertheless pulse contour analysis and impedance cardiography are known to provide only relative SV and CO values. Thus inert gas rebreathing gives us the possibility to calibrate these stroke volumes and cardiac outputs to absolute values. Success of this procedure was shown during former parabolic flights.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers (men or women)
* Aged from 18 to 55
* Affiliated to a Social Security System
* Who accepted to take part in the study
* Who have given their written stated consent
* Who already participated in parabolic flights or performed a centrifuge run up to 4 G with head movements without occurrence of serious nausea or vomiting or cardiovascular discomfort.
* Who has passed a medical examination similar to a standard aviation medical examination for private pilot aptitude (JAR FCL3 Class 2 medical examination). There will be no additional test performed for subject selection.

Exclusion Criteria:

* Person who took part in a previous biomedical research protocol, of which exclusion period is not terminated
* Pregnant women
* Medication with beta blockers, ACE inhibitors, calcium channel blockers or diuretics.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Estimated)
Dates: Start 2011-06; Primary Completion 2015-11 (Estimated)

PRIMARY OUTCOMES:
systolic finger blood pressure | baseline
Heart rate | baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Umr Ucbn/Inserm U1075 Comete, Caen, Basse-Normandie, France